CLINICAL TRIAL: NCT01659255
Title: An Open-label, Multi-Center, Non-Randomised Phase I Dose-Escalation Study to Investigate the Safety and Tolerability of ONO-4059 (ONO/GS-4059) Given as Monotherapy in Patients With Relapsed/Refractory Non-Hodgkin's Lymphoma (NHL) and Relapsed/Refractory Chronic Lymphocytic Leukaemia (CLL)
Brief Title: Study to Evaluate the Safety and Tolerability of Tirabrutinib (ONO/GS-4059) Given as Monotherapy in Participants With Relapsed/Refractory NHL and CLL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4059POE001; 2011-005033-39 (EudraCT Number)
Record Dates: First submitted 2012-07-06; First posted 2012-08-07 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Non Hodgkins Lymphoma; Chronic Lymphocytic Leukaemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, B-Cell | interventions — tirabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (17):
- Tirabrutinib 20 mg Once Daily (CLL) (Experimental): Participants with relapsed/refractory chronic lymphocytic leukaemia (CLL) received tirabrutinib 20 mg once daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 40 mg Once Daily (CLL) (Experimental): Participants with relapsed/refractory CLL received tirabrutinib 40 mg once daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 80 mg Once Daily (CLL) (Experimental): Participants with relapsed/refractory CLL received tirabrutinib 80 mg once daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 160 mg Once Daily (CLL) (Experimental): Participants with relapsed/refractory CLL received tirabrutinib 160 mg once daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 320 mg Once Daily (CLL) (Experimental): Participants with relapsed/refractory CLL received tirabrutinib 320 mg once daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 400 mg Once Daily (CLL) (Experimental): Participants with relapsed/refractory CLL received tirabrutinib 400 mg once daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 500 mg Once Daily (CLL) (Experimental): Participants with relapsed/refractory CLL received tirabrutinib 500 mg once daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 600 mg Once Daily (CLL) (Experimental): Participants with relapsed/refractory CLL received tirabrutinib 600 mg once daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 300 mg Twice Daily (CLL) (Experimental): Participants with relapsed/refractory CLL received tirabrutinib 300 mg twice daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 20 mg Once Daily (NHL) (Experimental): Participants with relapsed/refractory non-Hodgkin's lymphoma (NHL) received tirabrutinib 20 mg once daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 40 mg Once Daily (NHL) (Experimental): Participants with relapsed/refractory NHL received tirabrutinib 40 mg once daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 80 mg Once Daily (NHL) (Experimental): Participants with relapsed/refractory NHL received tirabrutinib 80 mg once daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 160 mg Once Daily (NHL) (Experimental): Participants with relapsed/refractory NHL received tirabrutinib 160 mg once daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 320 mg Once Daily (NHL) (Experimental): Participants with relapsed/refractory NHL received tirabrutinib 320 mg once daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 480 mg Once Daily (NHL) (Experimental): Participants with relapsed/refractory NHL received tirabrutinib 480 mg once daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 600 mg Once Daily (NHL) (Experimental): Participants with relapsed/refractory NHL received tirabrutinib 600 mg once daily.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib 240 mg Twice Daily (NHL) (Experimental): Participants with relapsed/refractory NHL received tirabrutinib 240 mg twice daily.
  Interventions: Drug: Tirabrutinib

INTERVENTIONS:
Drug: Tirabrutinib — Capsules administered orally
  Other Names: ONO/GS-4059

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of tirabrutinib (formerly ONO/GS-4059) given as monotherapy to participants with relapsed/refractory non-Hodgkin's lymphoma (NHL) and chronic lymphocytic leukemia (CLL).

ELIGIBILITY:
Key Inclusion Criteria:

1. Males or females with a confirmed diagnosis of and documented history of relapsed or refractory malignant disease (B-cell lymphoma and/or CLL) for which no therapy of curative or high priority exists and for whom treatment with a Btk inhibitor may be deemed appropriate.
2. Age ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.

Key Exclusion Criteria:

1. Central nervous system (CNS) lymphoma.
2. Women who are pregnant or lactating.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-08-17 (Actual); Primary Completion 2015-02-23 (Actual); Study Completion 2016-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- France (3):
  - CHRU - Hopital Claude HURIEZ, Lille
  - Centre hospitalier Lyon Sud, Lyon
  - CHU St Eloi, Montpellier
- United Kingdom (3):
  - University Hospital of Wales, Cardiff
  - Leicester Royal Infirmary, Leicester
  - Derriford Hospital, Plymouth

REFERENCES:
- [Result] Walter HS, Salles GA, Dyer MJ. New Agents to Treat Chronic Lymphocytic Leukemia. N Engl J Med. 2016 Jun 2;374(22):2185-6. doi: 10.1056/NEJMc1602674. No abstract available. PMID 27248633
- [Result] Walter HS, Rule SA, Dyer MJ, Karlin L, Jones C, Cazin B, Quittet P, Shah N, Hutchinson CV, Honda H, Duffy K, Birkett J, Jamieson V, Courtenay-Luck N, Yoshizawa T, Sharpe J, Ohno T, Abe S, Nishimura A, Cartron G, Morschhauser F, Fegan C, Salles G. A phase 1 clinical trial of the selective BTK inhibitor ONO/GS-4059 in relapsed and refractory mature B-cell malignancies. Blood. 2016 Jan 28;127(4):411-9. doi: 10.1182/blood-2015-08-664086. Epub 2015 Nov 5. PMID 26542378
- [Result] Fegan, C, Bagshawe J, Salles G, et al. The Bruton's tyrosine kinase (BTK) inhibitor ONO-4059: promising single agent activity and well tolerated in patients with high risk chronic lymphocytic leukaemia (CLL). Paper presented at: 56th American Society of Hematology Annual Meeting and Exposition; December 6-9, 2014; San Franscisco, CA.
- [Result] Morschhauser F, Terriou L, Dyer M, et al. The Bruton's tyrosine kinase (BTK) inhibitor ONO-4059: promising single agent activity in patients with relapsed and refractory NHL. Haematologica. 2014 Jun; 99: 150.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe. The first participant was screened on 17 August 2012. The last study visit occurred on 11 January 2016.
Pre-assignment Details: 102 participants were screened.
Period: Overall Study
Arm/Group | Tirabrutinib 20 mg Once Daily (CLL) | Tirabrutinib 40 mg Once Daily (CLL) | Tirabrutinib 80 mg Once Daily (CLL) | Tirabrutinib 160 mg Once Daily (CLL) | Tirabrutinib 320 mg Once Daily (CLL) | Tirabrutinib 400 mg Once Daily (CLL) | Tirabrutinib 500 mg Once Daily (CLL) | Tirabrutinib 600 mg Once Daily (CLL) | Tirabrutinib 300 mg Twice Daily (CLL) | Tirabrutinib 20 mg Once Daily (NHL) | Tirabrutinib 40 mg Once Daily (NHL) | Tirabrutinib 80 mg Once Daily (NHL) | Tirabrutinib 160 mg Once Daily (NHL) | Tirabrutinib 320 mg Once Daily (NHL) | Tirabrutinib 480 mg Once Daily (NHL) | Tirabrutinib 600 mg Once Daily (NHL) | Tirabrutinib 240 mg Twice Daily (NHL)
Started | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 5 | 8 | 21 | 10 | 9 | 3
Completed | 1 | 2 | 4 | 3 | 3 | 2 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 3 | 2 | 4 | 0
Not Completed | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 3 | 3 | 4 | 8 | 18 | 8 | 5 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0
Not completed — Progressive Disease | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 3 | 5 | 13 | 6 | 2 | 3
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Investigator Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Sponsor's Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Completed Treatment Per Protocol at the Time | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Participant Went on to Have an Allograft | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all the participants who received at least 1 dose of study drug.
Groups:
- Tirabrutinib 20 mg Once Daily (CLL): Participants with relapsed/refractory CLL received tirabrutinib 20 mg once daily.
- Tirabrutinib 20 mg Once Daily (NHL): Participants with relapsed/refractory NHL received tirabrutinib 20 mg once daily.
- Total: Total of all reporting groups
Arm/Group | Tirabrutinib 20 mg Once Daily (CLL) | Tirabrutinib 40 mg Once Daily (CLL) | Tirabrutinib 80 mg Once Daily (CLL) | Tirabrutinib 160 mg Once Daily (CLL) | Tirabrutinib 320 mg Once Daily (CLL) | Tirabrutinib 400 mg Once Daily (CLL) | Tirabrutinib 500 mg Once Daily (CLL) | Tirabrutinib 600 mg Once Daily (CLL) | Tirabrutinib 300 mg Twice Daily (CLL) | Tirabrutinib 20 mg Once Daily (NHL) | Tirabrutinib 40 mg Once Daily (NHL) | Tirabrutinib 80 mg Once Daily (NHL) | Tirabrutinib 160 mg Once Daily (NHL) | Tirabrutinib 320 mg Once Daily (NHL) | Tirabrutinib 480 mg Once Daily (NHL) | Tirabrutinib 600 mg Once Daily (NHL) | Tirabrutinib 240 mg Twice Daily (NHL) | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 5 | 8 | 21 | 10 | 9 | 3 | 90
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 1 | 0 | 3 | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 2 | 3 | 7 | 7 | 6 | 2 | 1 | 39
  ≥ 65 years | 2 | 3 | 1 | 2 | 2 | 1 | 1 | 2 | 3 | 3 | 1 | 2 | 1 | 14 | 4 | 7 | 2 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 8 | 3 | 3 | 2 | 25
  Male | 3 | 3 | 3 | 2 | 2 | 3 | 3 | 2 | 2 | 1 | 2 | 5 | 7 | 13 | 7 | 6 | 1 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 3 | 4 | 1 | 3 | 3 | 2 | 3 | 2 | 3 | 3 | 3 | 7 | 16 | 9 | 8 | 3 | 75
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Other | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 4 | 1 | 0 | 0 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Dose-Limiting Toxicities
Description: Dose Limiting Toxicities (DLT) were defined as follows:
  * All Common Terminology Criteria (CTC) Grade 4 tirabrutinib related adverse events
  * All CTC Grade 3 tirabrutinib related adverse events, with the exception of the following:
    * CTC Grade 3 lymphocytosis considered an expected outcome of therapy
  Any toxicity which in the opinion of the Investigator is attributed to a participant's underlying disease was not considered a DLT.
Time Frame: Day 1 through Day 28
Population: The Safety Analysis Set included all the participants who received at least 1 dose of study drug. Per planned analysis, data for DLTs were summarized by dose level received by participants with NHL and CLL.
Measure: Number; unit: percentage of participants
Arm/Group | Tirabrutinib 20 mg Once Daily (CLL) | Tirabrutinib 40 mg Once Daily (CLL) | Tirabrutinib 80 mg Once Daily (CLL) | Tirabrutinib 160 mg Once Daily (CLL) | Tirabrutinib 320 mg Once Daily (CLL) | Tirabrutinib 400 mg Once Daily (CLL) | Tirabrutinib 500 mg Once Daily (CLL) | Tirabrutinib 600 mg Once Daily (CLL) | Tirabrutinib 300 mg Twice Daily (CLL) | Tirabrutinib 20 mg Once Daily (NHL) | Tirabrutinib 40 mg Once Daily (NHL) | Tirabrutinib 80 mg Once Daily (NHL) | Tirabrutinib 160 mg Once Daily (NHL) | Tirabrutinib 320 mg Once Daily (NHL) | Tirabrutinib 480 mg Once Daily (NHL) | Tirabrutinib 600 mg Once Daily (NHL) | Tirabrutinib 240 mg Twice Daily (NHL)
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 5 | 8 | 21 | 10 | 9 | 3
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 33.3 | 0.0 | 0.0 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 4.8 | 10.0 | 22.2 | 0.0

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate (ORR) was defined as the percentage of participants who achieve a best overall response of complete remission (CR, unconfirmed complete response (CRu), complete response with incomplete marrow recovery (CRi)) or partial remission (PR, nodal PR) during study as assessed by the investigator.
  ORR assessment was defined per following standardized criteria:
  * NHL: Cheson, 1999
  * CLL: International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008
Time Frame: Up to Cycle 37 (28 days for each cycle) plus 6-month intervals thereafter until disease progression (maximum: up to 39 months)
Population: The Full Analysis Set included all the participants who received at least 1 dose of study drug. Per planned analysis, data for overall response rate were summarized by overall CLL group and NHL subgroup.
Measure: Number; unit: percentage of participants
Groups:
- Chronic Lymphocytic Leukaemia: Participants with relapsed/refractory CLL received tirabrutinib until disease progression or until the participant entered into a possible future tirabrutinib study.
- NHL Subtype FL: Participants with NHL subtype follicular lymphoma (FL) received tirabrutinib until disease progression or until the participant entered into a possible future tirabrutinib study.
- NHL Subtype SLL: Participants with NHL subtype small lymphocytic lymphoma (SLL) received tirabrutinib until disease progression or until the participant entered into a possible future tirabrutinib study.
- NHL Subtype WM: Participants with NHL subtype Waldenstrom macroglobulinemia (WM) received tirabrutinib until disease progression or until the participant entered into a possible future tirabrutinib study.
- NHL Subtype MZL: Participants with NHL subtype marginal zone lymphoma (MZL) received tirabrutinib until disease progression or until the participant entered into a possible future tirabrutinib study.
- NHL Subtype DLBCL: Participants with NHL subtype diffuse large B-cell lymphoma (DLBCL) received tirabrutinib until disease progression or until the participant entered into a possible future tirabrutinib study.
- NHL Subtype MCL: Participants with NHL subtype mantle cell lymphoma (MCL) received tirabrutinib until disease progression or until the participant entered into a possible future tirabrutinib study.
Arm/Group | Chronic Lymphocytic Leukaemia | NHL Subtype FL | NHL Subtype SLL | NHL Subtype WM | NHL Subtype MZL | NHL Subtype DLBCL | NHL Subtype MCL
Number analyzed (Participants) | 28 | 5 | 1 | 3 | 2 | 35 | 16
percentage of participants | 85.7 | 0.0 | 0.0 | 33.3 | 50.0 | 31.4 | 68.8

3. Secondary Outcome: Pharmacokinetic (PK) Parameter: Cmax of Tirabrutinib
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: Pre-dose, then 30 minutes, 1, 2, 3, 4, 6, 8, 12 hours post-dose at Cycle 1, Day 28
Population: Participants in the PK Analysis Set (all participants who received at least 1 dose of study drug and had at least 1 nonmissing postdose concentration value for the corresponding analyte in plasma) with available data were analyzed. Per planned analysis, data for PK parameters were summarized by dose cohorts.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Tirabrutinib 20 mg Once Daily (CLL or NHL): Participants with relapsed/refractory CLL or NHL received tirabrutinib 20 mg once daily.
- Tirabrutinib 40 mg Once Daily (CLL or NHL): Participants with relapsed/refractory CLL or NHL received tirabrutinib 40 mg once daily.
- Tirabrutinib 80 mg Once Daily (CLL or NHL): Participants with relapsed/refractory CLL or NHL received tirabrutinib 80 mg once daily.
- Tirabrutinib 160 mg Once Daily (CLL or NHL): Participants with relapsed/refractory CLL or NHL received tirabrutinib 160 mg once daily.
- Tirabrutinib 320 mg Once Daily (CLL or NHL): Participants with relapsed/refractory CLL or NHL received tirabrutinib 320 mg once daily.
- Tirabrutinib 600 mg Once Daily (CLL or NHL): Participants with relapsed/refractory CLL or NHL received tirabrutinib 600 mg once daily.
Arm/Group | Tirabrutinib 20 mg Once Daily (CLL or NHL) | Tirabrutinib 40 mg Once Daily (CLL or NHL) | Tirabrutinib 80 mg Once Daily (CLL or NHL) | Tirabrutinib 160 mg Once Daily (CLL or NHL) | Tirabrutinib 320 mg Once Daily (CLL or NHL) | Tirabrutinib 400 mg Once Daily (CLL) | Tirabrutinib 480 mg Once Daily (NHL) | Tirabrutinib 500 mg Once Daily (CLL) | Tirabrutinib 600 mg Once Daily (CLL or NHL) | Tirabrutinib 240 mg Twice Daily (NHL) | Tirabrutinib 300 mg Twice Daily (CLL)
Number analyzed (Participants) | 6 | 6 | 5 | 10 | 17 | 2 | 7 | 3 | 6 | 3 | 3
ng/mL | 73.4 (18.26) | 164.5 (47.22) | 241 (90.68) | 539.6 (141.58) | 1181.6 (380.39) | 826.5 (499.92) | 1240.3 (516.99) | 1230 (285.83) | 1265.2 (486.21) | 704.3 (254.51) | 674.3 (93.78)

4. Secondary Outcome: PK Parameter: AUCtau of Tirabrutinib
Description: AUCtau is defined as concentration of drug over dosing interval.
Time Frame: Pre-dose, then 30 minutes, 1, 2, 3, 4, 6, 8, 12 hours post-dose at Cycle 1, Day 28
Population: Participants in the PK Analysis Set with available data were analyzed. Per planned analysis, data for PK parameters were summarized by dose cohorts.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Tirabrutinib 20 mg Once Daily (CLL or NHL) | Tirabrutinib 40 mg Once Daily (CLL or NHL) | Tirabrutinib 80 mg Once Daily (CLL or NHL) | Tirabrutinib 160 mg Once Daily (CLL or NHL) | Tirabrutinib 320 mg Once Daily (CLL or NHL) | Tirabrutinib 400 mg Once Daily (CLL) | Tirabrutinib 480 mg Once Daily (NHL) | Tirabrutinib 500 mg Once Daily (CLL) | Tirabrutinib 600 mg Once Daily (CLL or NHL) | Tirabrutinib 240 mg Twice Daily (NHL) | Tirabrutinib 300 mg Twice Daily (CLL)
Number analyzed (Participants) | 6 | 6 | 5 | 10 | 17 | 2 | 7 | 3 | 5 | 3 | 2
h*ng/mL | 306.4 (74.92) | 660.1 (310.95) | 762 (374.94) | 2681.8 (1055.17) | 5664.8 (1829.07) | 5259.5 (3166.57) | 7999.8 (2006.19) | 6766.9 (1025.64) | 8442.2 (2499.22) | 3415.5 (1296.47) | 3297.2 (1330)

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to the last dose date plus 30 days (maximum: 36 months); All-Cause Mortality: First dose date up to 39 months
Description: The Safety Analysis Set included all the participants who received at least 1 dose of study drug. Per planned analysis, data were summarized by overall groups for NHL and CLL pooling all participants regardless of dose level received.
Groups:
- Non-Hodgkin's Lymphoma: Participants with relapsed/refractory NHL received tirabrutinib until disease progression or until the participant entered into a possible future tirabrutinib study.
Arm/Group | Chronic Lymphocytic Leukaemia | Non-Hodgkin's Lymphoma
All-Cause Mortality (participants affected / at risk) | 5/28 | 38/62
Serious Adverse Events (participants affected / at risk) | 17/28 | 23/62
Other Adverse Events (participants affected / at risk) | 28/28 | 55/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Lymphocytic Leukaemia (N=28) | Non-Hodgkin's Lymphoma (N=62)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Lymphocytic infiltration (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 1
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Adverse drug reaction (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Ill-defined disorder (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 1
Ear infection (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
H1n1 influenza (Infections and infestations) | 0 | 1
Hepatitis E (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster oticus (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 4 | 3
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 2 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 1 | 2
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Myeloma cast nephropathy (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Lymphocytic Leukaemia (N=28) | Non-Hodgkin's Lymphoma (N=62)
Anaemia (Blood and lymphatic system disorders) | 9 | 23
Leukopenia (Blood and lymphatic system disorders) | 2 | 2
Lymphopenia (Blood and lymphatic system disorders) | 2 | 12
Neutropenia (Blood and lymphatic system disorders) | 9 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 18
Ear pain (Ear and labyrinth disorders) | 3 | 0
Conjunctival haemorrhage (Eye disorders) | 2 | 1
Eye haemorrhage (Eye disorders) | 3 | 0
Eye pruritus (Eye disorders) | 2 | 2
Glaucoma (Eye disorders) | 2 | 0
Ocular hyperaemia (Eye disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 8
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 18
Dry mouth (Gastrointestinal disorders) | 2 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 12
Vomiting (Gastrointestinal disorders) | 5 | 9
Asthenia (General disorders) | 3 | 9
Fatigue (General disorders) | 5 | 7
Oedema peripheral (General disorders) | 2 | 8
Pyrexia (General disorders) | 7 | 7
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Hypogammaglobulinaemia (Immune system disorders) | 2 | 0
Bronchitis (Infections and infestations) | 3 | 4
Cellulitis (Infections and infestations) | 3 | 0
Chronic sinusitis (Infections and infestations) | 2 | 0
Ear infection (Infections and infestations) | 2 | 1
Eye infection (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 4 | 3
Influenza (Infections and infestations) | 2 | 2
Laryngitis (Infections and infestations) | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 5 | 6
Lung infection (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 9 | 11
Oral herpes (Infections and infestations) | 3 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 2 | 8
Sinobronchitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 5
Urinary tract infection (Infections and infestations) | 3 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 10 | 8
Fall (Injury, poisoning and procedural complications) | 8 | 5
Laceration (Injury, poisoning and procedural complications) | 4 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 3 | 1
Blood bilirubin increased (Investigations) | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 5
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 3 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Carpal tunnel syndrome (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 4 | 1
Dysaesthesia (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 4 | 5
Paraesthesia (Nervous system disorders) | 4 | 0
Anxiety (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 2 | 5
Prostatomegaly (Reproductive system and breast disorders) | 2 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Acne (Skin and subcutaneous tissue disorders) | 3 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 3
Eczema (Skin and subcutaneous tissue disorders) | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 5 | 2
Macule (Skin and subcutaneous tissue disorders) | 6 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 6 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 5
Purpura (Skin and subcutaneous tissue disorders) | 5 | 6
Rash macular (Skin and subcutaneous tissue disorders) | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 2
Swelling face (Skin and subcutaneous tissue disorders) | 2 | 1
Haematoma (Vascular disorders) | 7 | 3
Hypertension (Vascular disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years